CLINICAL TRIAL: NCT05717699
Title: Oncolytic Virus Ad-TD-nsIL12 for Progressive Pediatric Diffuse Intrinsic Pontine Glioma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Hongwei Zhang, Professor, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ad-TD-nsIL12 for Pro-DIPG
Record Dates: First submitted 2022-12-18; First posted 2023-02-08 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Oncolytic Virus; Diffuse Intrinsic Pontine Glioma; Adverse Drug Event
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Multiple intratumoral injections of Ad-TD-nsIL12.
  Interventions: Biological: Ad-TD-nsIL12

INTERVENTIONS:
Biological: Ad-TD-nsIL12 — After stereotactic biopsy, the Ommaya reservoir will be inserted through the biopsy channel and two injections of Ad-TD-nsIL12 will be delivered after surgery by Ommaya reservoir (with an interval of 3days). The interval between following injections in the subsequent treatment period will be 3 weeks ±4 days. The assigned dose for each patient will be 3x10^9vp, 1x10^10vp or 3x10^10 vp suspended in 1 ml NS according to cohort design.

SUMMARY:
This is a single-arm, single-center, drug safety assessment clinical trial with a 3+3 dose escalation design, to observe the safety, tolerability and toxicity of a novel oncolytic virus Ad-TD-nsIL12 intratumoral injection in progressive DIPG patients (NCI-CTCAE V5.0).

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent of the parents or patient.
2. After surgical resection, biopsy, chemotherapy, or radiation therapy, tumor progression must be confirmed by MRI scan.
3. Biopsy is performed prior to injection of Ad-TD-nsIL12 to confirm DIPG (frozen section-based).
4. Pre-enrollment patients LPS (patients aged ≥1 and <16 years) and KPS (patients aged ≥16 years) ≥ 50.
5. Patient must be, in the investigator opinion, able to comply with all the protocol procedures.
6. Age 1-18 years.
7. A negative pregnancy test in fertile women (women are considered of childbearing potential (WOCBP) after menarche, unless permanently infertile, including hysterectomy, bilateral salpingectomy, and bilateral oophorectomy).
8. Lesion considered by the investigator to be accessible for stereotactic biopsy.

Exclusion Criteria:

1. Serious infections or intercurrent conditions, including but not limited to severe renal failure, liver failure, heart failure, or bone marrow failure, which are not permitted for inclusion according to the investigator's criteria. Patients must be afebrile (<38℃) at the time of viral therapy.
2. Other investigational medications within 30 days prior to viral treatment.
3. Participants with immunodeficiency, autoimmune disease, or active hepatitis.
4. Any medical or psychological condition that might interfere with the patient's ability to participate if older than 16 years or parents ability when younger than 16, or give informed consent or would compromise the patient's ability to tolerate therapy or any disease that will obscure toxicity or dangerously alter drug metabolism.
5. Tumor with multiple location.
6. Pregnant or breast-feeding females.
7. Severe bone marrow hypoplasia.
8. Transaminases (aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT)) or total bilirubin > 3 times the upper limit of normal.
9. Neutrophils < 1x10^9/L.
10. Platelets ≤ 100x10^9/L.
11. Hemoglobin < 9g/dl.
12. Patients with Li-Fraumini syndrome or a known germline defect in the retinoblastoma gene or its associated pathways.
13. Administer any type of vaccine within 30 days prior to Ad-TD-nsIL12 administration.
14. Blood transfusions or drugs (such as G-CSF) within 28 days before viral treatment to treat pancytopenia or other hematological disorders.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2025-01-04 (Estimated); Study Completion 2028-01-04 (Estimated)

PRIMARY OUTCOMES:
Safety of Ad-TD-nsIL12 intratumoral injection in progressive pediatric DIPG patients. | 3 months after virus injection
  The trial will look for possible hematologic and neurologic toxicity of Ad-TD-nsIL12 by NCI-CTCAE v5.0 to determine maximum tolerated dose of this oncolytic adenovirus.

SECONDARY OUTCOMES:
Tumor response | 3 months after virus injection
  To determine tumor response by RAPNO criteria
Over-all survival | 12 months after virus injection
  To determine overall survival at 12 months (OS12).
QoL | 2 years after virus injection
  To measure quality of life baseline assessment and any changes over time by PedsQLTM criteria.
Sample Collection | 3 months after virus injection
  Pre- and post- treatment tumor tissue will be collected and tested to determine the immune response of patients. Collected blood will be used to test possible hematotoxicity of Ad-TD-nsIL12.

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Zhang, Prof., Principal Investigator — Capital Medical University
Locations (1):
- Sanbo Brain Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Zhang Z, Zhang C, Miao J, Wang Z, Wang Z, Cheng Z, Wang P, Dunmall LSC, Lemoine NR, Wang Y. A Tumor-Targeted Replicating Oncolytic Adenovirus Ad-TD-nsIL12 as a Promising Therapeutic Agent for Human Esophageal Squamous Cell Carcinoma. Cells. 2020 Nov 10;9(11):2438. doi: 10.3390/cells9112438. PMID 33182528
- [Background] Bortolanza S, Bunuales M, Otano I, Gonzalez-Aseguinolaza G, Ortiz-de-Solorzano C, Perez D, Prieto J, Hernandez-Alcoceba R. Treatment of pancreatic cancer with an oncolytic adenovirus expressing interleukin-12 in Syrian hamsters. Mol Ther. 2009 Apr;17(4):614-22. doi: 10.1038/mt.2009.9. Epub 2009 Feb 17. PMID 19223865
- [Background] Wang P, Li X, Wang J, Gao D, Li Y, Li H, Chu Y, Zhang Z, Liu H, Jiang G, Cheng Z, Wang S, Dong J, Feng B, Chard LS, Lemoine NR, Wang Y. Re-designing Interleukin-12 to enhance its safety and potential as an anti-tumor immunotherapeutic agent. Nat Commun. 2017 Nov 9;8(1):1395. doi: 10.1038/s41467-017-01385-8. PMID 29123084